CLINICAL TRIAL: NCT01622452
Title: Neurocognitive Deficits Related to Cardiac Surgery Intervention With Extracorporeal Circulation. Correlations Between Neuropsychological Tests and Functional MRI Techniques (Spectroscopy, Diffusion and Morphometry)
Brief Title: Post Cardiac Surgery Neurocognitive Decline: Correlations Between Neuropsychological Tests and Functional MRI Techniques
Acronym: CardChNeuroMRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Responsible Party: Principal Investigator, Montanaro Domenico, Responsible of the Neuroradiological Unit, Foundation CNR - Regione Toscana G. Monasterio, Fondazione Toscana Gabriele Monasterio
Other Study IDs: 396/12 FTGM
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative cognitive dysfunction; Cognitive decline; Valve surgery; Cardiac surgery; Diffusion Tensor Imaging; Brain Morphometry; 1H-Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative cognitive decline (POCD) is a frequent complication after cardiac surgery. It is estimated that 40-70% of all cardiac patients show cognitive dysfunction during the first post-surgical week. Six weeks after surgery, this incidence decreases to 10-40% and the figure remains stable over the long-term.

The investigators will recruit 50 patients undergoing elective valve surgery and each patient will receive complete evaluation a) preoperative, one week before surgery; b) early postoperative, before hospital discharge; and c) late postoperative, 8 weeks follow up.

The investigators will apply Diffusion Tensor Imaging, 1Proton-Magnetic Resonance Spectroscopy and Morphometry studies with correlation to neuropsychological test battery to evaluate POCD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective valve surgery in Ospedale del Cuore, Fondazione G. Monasterio, Massa, Italy will prospectively enter the study.

Exclusion Criteria:

* History of head trauma, seizures, stroke, carotid artery stenosis (>70%)
* History of any major surgery with general anesthesia
* Preoperative MMSE score less than 23 to exclude patients with dementia and mild cognitive impairment (MCI)
* Subjects who will be unable to complete the baseline neuropsychological battery due to cognitive impairment, psychiatric disease, substance abuse, blindness, or poor knowledge of Italian language
* Any major neurological complication after CABG surgery (stroke, seizures, encephalopathy not resolving within few postoperative days)
* if any contraindications to MRI safety, indicated in local MRI safety protocol

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective valve surgery in Ospedale del Cuore, Fondazione G. Monasterio, Massa, Italy and matching inclusion/exclusion criteria will prospectively enter the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Brain MRI microstructural/functional alteration due to cardiac surgery in association with POCD | 32 months
  On the basis of scientific literature, the patients during the first post-cardiosurgical week can show cognitive dysfunction in 40-70% of the cases, decreasing after 6 weeks to 10-40%, remaining stable over the long-term. To identify corresponding brain specific microstructural variations, simultaneously to the neuropsychological evaluation, the same group of patients will undergo to MRI with standard sequence and advanced morpho-structural methods (DTI and VBM). Comparing data with a group of healthy age-matched subjects (20), quantitative measurements by VBM and DTI will be carried out to identify GM and WM variations, subsequently correlated with onset of POCD.
Brain MRI metabolic alteration due to cardiac surgery in association with POCD | 32 months
  To explore pre- and post- operative metabolic changes on the brain using in-vivo proton magnetic resonance spectroscopy (1H-MRS) after otherwise successful cardiac surgery with no major neurological event.